CLINICAL TRIAL: NCT04138121
Title: Impact of Change of Head and Neck Position on Cricothyroid Membrane Localization and Membrane Height in Parturient Patients: an Observational Study
Brief Title: Impact of Change of Head and Neck Position on Cricothyroid Membrane Localization and Membrane Height in Parturient Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-05
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Airway Complication of Anesthesia
Keywords: cricothyroid membrane; pregnancy; ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Experimental): Ultrasound measurements of the cricothyroid membrane.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound scan of the cricothyroid membrane

SUMMARY:
The cricothyroid membrane acts a route through which the upper airway can be accessed in order to provide oxygen and ventilation to patients. The need to provide oxygen and ventilation to patients is essential particularly under general anesthesia, where patients may lose the ability to breathe for themselves. Access through this membrane to provide oxygen and ventilation is critical in emergency situations where other traditional means to access the airway (e.g through endotracheal ventilation, supraglottic airway devices or face mask ventilation) have failed. It is known that due to the physiological changes of pregnancy, the upper airway of the body undergoes changes that can make accessing the airway through traditional means more difficult. Ultrasound is becoming increasingly popular due to its ability to identify the cricothyroid membrane, to improve success in accessing the airway through the cricothyroid membrane. Studies to date in non pregnant adults have shown that alterations in the head and neck position can alter the position and size of the cricothyroid membrane. No study to date however has looked at how changing the position of the head and neck effects the position and size of the cricothyroid membrane in pregnant patients. It is important to study these changes in the pregnant population, given the physiological changes of pregnancy that make accessing the airway through traditional methods more difficult in non pregnant patients. The investigators hypothesize that in pregnant patients in the third trimester, that changing the head from the neutral to maximally extended neck position will alter the position of the cricothyroid membrane in relation to anatomical skin markings between positions. The investigators also hypothesize that in pregnant patients in the third trimester that changing the head from the neutral to maximally extended neck position will increase the size of the cricothyroid membrane. The investigatorsalso aim to determine at what position in the neck a theoretical standardized incision will allow access to the cricothyroid membrane.

DETAILED DESCRIPTION:
This is an observational study.

Participants:

1. One of two anesthesiologists trained in cricothyroid membrane ultrasound scanning technique in pregnant population (study investigators)
2. Subjects to be assessed: pregnant patients in their third trimester on the labor and delivery floor comfortable enough to take part in the study

Two anesthesiologists will undergo ultrasound imaging training by an expert staff anesthesiologist whom is already trained in the procedure. As per previous published evidence on this, the investigator will need to correctly identify the location of cricothyroid membrane and its height in 15 volunteers. This will constitute the standardized training component of the study.

Upon admission to the Labor and Delivery floor, women will be further explained the protocol and asked to sign the consent form. Then, they will have the cricothyroid membrane assessed, as per description above, and quantitative assessment will be performed. Firstly, quantitative assessment of the height of the cricothyroid membrane will be performed in the supine position (with left uterine displacement) with the neck in the neutral position. The central point of the cricothyroid membrane will be marked using a removable skin ink marker. The patient will then be asked to fully their neck. The change in distance of the midpoint of the cricothyroid membrane from the neutral head and neck position to fully extended positioned will be performed, as will the change in height of the cricothyroid membrane between the two positions.

Quantitative assessment for change in central cricothyroid membrane distance will be done with measuring central points marked on the patients neck with skin marker ink. Quantitative assessment of change in cricoid thyroid membrane will be conducted using caliper measuring software build into the ultrasound machinery. Finally, the investigators will establish the starting distance above the sternal notch over which a theoretical 8cm incision in the neck which will overlie the cricothyroid membrane. This will be done by measuring the distance above the sternal notch with a surgical measuring ruler.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients in third trimester (>28/40 weeks)
* Ability to understand the rationale of the study assessments and to provide signed consent.

Exclusion Criteria:

* Neck arthritis
* Cervical stenosis
* Known cervical degenerative disc disease
* Rheumatoid Arthritis
* Any restriction of neck movement
* Upper limb neurology
* Patient refusal
* Non pregnant patients
* Pregnant patients less than 28 weeks pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Cricothyroid membrane position change | 30 minutes
  To measure the distance the center of the cricothyroid membrane changes position on ultrasound between neutral and maximal neck extension in third trimester patients.

SECONDARY OUTCOMES:
Cricothyroid membrane size change | 30 minutes
  To measure the distance that the size of the cricothyroid membrane changes position on ultrasound between neutral and maximal neck extension in third trimester patients.
Distance above sternal notch | 30 minutes
  The starting distance above the sternal notch in the neck over which an 8cm incision in the neck should overlie the cricothyroid membrane

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No